CLINICAL TRIAL: NCT00357877
Title: Prevention of Adult Caries Study
Brief Title: Prevention of Adult Caries Study (PACS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DE017753-01; U01DE017753 (NIH)
Record Dates: First submitted 2006-07-26; First posted 2006-07-28 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Caries, Dental
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Dental Coating (Placebo Comparator): Dental coating with all ingredients except Chlorhexidine topically applied by dental professional supragingivally to the full dentition
  Interventions: Other: Placebo
- Active Dental Coating (Active Comparator): 10% w/v chlorhexidine acetate coating FDA IND #45466. Dental coating with all ingredients including Chlorhexidine topically applied by dental professional supragingivally to the full dentition
  Interventions: Drug: 10% w/v chlorhexidine acetate coating FDA IND #45466

INTERVENTIONS:
Drug: 10% w/v chlorhexidine acetate coating FDA IND #45466 — Dental coating topically applied by dental professional supragingivally to the full dentition
  Other Names: CHX
  Arms: Active Dental Coating
Other: Placebo
  Arms: Placebo Dental Coating

SUMMARY:
Adult tooth decay is an infectious disease that afflicts the majority of Americans aged 55 and older and is the most common chronic disease at midlife with an ever growing economic toll. Despite the fact that specific bacteria cause tooth decay, no FDA-approved anti-microbial treatment for decay is available to the American dental professional. The Prevention of Adult Caries Study (PACS) is a study designed to evaluate the efficacy of a topical, temporary, 10% w/v chlorhexidine dental coating in reducing new decay in adult dental patients at risk for decay.

DETAILED DESCRIPTION:
The Prevention of Adult Caries Study (PACS) is a randomized, double-blind, placebo-controlled Phase III clinical trial conducted under F.D.A. Investigational New Drug license #45,466, with a target enrollment of 1000 at four clinical centers with vastly different populations. The centers participating in this proposed research are: Kaiser Permanente's Dental Plan in Portland, Oregon; Tufts University Dental Clinic in central Boston, Massachusetts; Delta Dental Massachusetts' Dental Clinic in Southborough, Massachusetts; and the dental clinic of the Tuba City Regional Health Care Corporation in Tuba City, Arizona. Kaiser Permanente's Center for Health Research in Portland, Oregon will act as the data-coordinating center, and Tufts University will act as the Administrative Center. This study is designed to evaluate the efficacy of a topical, temporary, 10% w/v chlorhexidine dental coating in reducing caries increment in at-risk adult dental patients. This study will treat participants in months 1(4 weekly applications) and 7(1 application) with final outcome measured at 13 months after randomization. Examiners were trained and certified before data collection started and were recalibrated annually. The primary outcome analysis in the intent -to- treat sample compares active to placebo group on the rank-normalized caries increment score, adjusting for examiner, age and age squared. Multiple imputation (data augmentation using MCMC) will be used to replace missing outcome. Planned secondary analysis examine the secondary caries increment outcomes using the same model, as well as parallel analyses in the per-protocol group. Safety of the coating will be evaluated by comparing development of resistant S. mutans or C. albicans as well as incidence of MedDRA-coded adverse events between the two arms.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* at least 20 intact natural teeth, excluding third molars
* 2 or more lesions, of which at least one must be a cavitated D2 or D3
* willing and able to provide informed consent

Exclusion Criteria

* pregnant or planning to become pregnant or planning to become pregnant during the study (breastfeeding is permitted)
* use of fixed orthodontic appliances
* allergic to any of the ingredients of the study medication
* long-term antibiotic therapy
* a history of, or currently active, radiation therapy for cancers of the head or neck
* Sjögren's syndrome
* advanced periodontitis
* consumption of the equivalent of more than five servings of acidic or sugared drinks per day
* having 10 or more lesions requiring restorative care at the time of the screening visit
* remineralization therapy within one month of randomization
* investigator discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 983 (Actual)
Dates: Start 2006-07; Primary Completion 2009-08 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Athena Papas, PhD DMD, Principal Investigator — Tufts University of Dental Medicine
Locations (4):
- United States (4):
  - Tuba City Regional Health Care, Tuba City, Arizona
  - Tufts University School of Dental Medicine, Boston, Massachusetts
  - Dental Services of Massachusetts, Boston, Massachusetts
  - Center for Health Research, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Papas AS, Vollmer WM, Gullion CM, Bader J, Laws R, Fellows J, Hollis JF, Maupome G, Singh ML, Snyder J, Blanchard P; PACS Collaborative Group. Efficacy of chlorhexidine varnish for the prevention of adult caries: a randomized trial. J Dent Res. 2012 Feb;91(2):150-5. doi: 10.1177/0022034511424154. Epub 2011 Dec 7. PMID 22156917
- [Derived] Singh M, Papas A, Vollmer W, Bader J, Laws R, Maupome G, Snyder J, Blanchard P. Predictors of coronal caries progression in adults: results from the Prevention of Adult Caries Study. Community Dent Oral Epidemiol. 2013 Dec;41(6):558-64. doi: 10.1111/cdoe.12059. Epub 2013 Jul 9. PMID 23834229
- [Derived] Banting DW, Amaechi BT, Bader JD, Blanchard P, Gilbert GH, Gullion CM, Holland JC, Makhija SK, Papas A, Ritter AV, Singh ML, Vollmer WM. Examiner training and reliability in two randomized clinical trials of adult dental caries. J Public Health Dent. 2011 Fall;71(4):335-44. doi: 10.1111/j.1752-7325.2011.00278.x. Epub 2011 Aug 17. PMID 22320292
- [Derived] Vollmer WM, Papas AS, Bader JD, Maupome G, Gullion CM, Hollis JF, Snyder JJ, Fellows JL, Laws RL, White BA; PACS Collaborative Research Group. Design of the Prevention of Adult Caries Study (PACS): a randomized clinical trial assessing the effect of a chlorhexidine dental coating for the prevention of adult caries. BMC Oral Health. 2010 Oct 5;10:23. doi: 10.1186/1472-6831-10-23. PMID 20923557

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Dental Coating (CHX): Dental coating with all ingredients including Chlorhexidine topically applied by dental professional supragingivally to the full dentition. 10% w/v chlorhexidine acetate coating FDA IND #45466.
Period: Overall Study
Arm/Group | Placebo Dental Coating | Active Dental Coating (CHX)
Started | 493 | 490
Completed | 467 | 460
Not Completed | 26 | 30
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 20 | 23
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Administrative withdrawal | 1 | 1
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Active Dental Coating: Dental coating with all ingredients including Chlorhexidine topically applied by dental professional supragingivally to the full dentition
- Total: Total of all reporting groups
Arm/Group | Placebo Dental Coating | Active Dental Coating | Total
Number analyzed (Participants) | 493 | 490 | 983
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 463 | 459 | 922
  >=65 years | 30 | 31 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (14.3) | 42.9 (14.3) | 42.8 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 242 | 250 | 492
  Male | 251 | 240 | 491
Region of Enrollment [Number; unit: participants]
  United States | 493 | 490 | 983

OUTCOME MEASURES:

1. Primary Outcome: Total Net D12FS Caries Increment (Total of Non-cavitated Lesions (D1), Cavitated Lesions (D2) and Sound Surfaces (S))
Description: Study duration was too short to have progression from D2 (cavitated lesions) to D3 (cavitated lesions that involved dentin). D2 and D3 were treated equivalently for analysis.
  This measure is computed as the sum of weighted counts of transitions in tooth surface status (root and coronal surfaces combined) from randomization to the 13-month follow-up visit. Disease progression had a positive weight (e.g., S-to-D1 (sound to non-cavitated lesion) or D1-to-D2 (non-cavitated to cavitated lesion) = 1, S-to-D2 (sound to cavitated lesion)= 2). Reversal had a negative weight (e.g., D1-to-S = -1). No change, transitions to or from missing or unscorable, and impossible transitions had 0 weight. Incident fillings and crowns were treated the same as incident D2 lesions for purposes of scoring. More details of the transition weights may be found at Vollmer WM et al. (2010). Design of the Prevention of Adult Caries Study (PACS): a randomized clinical trial assessing the effect of a
Time Frame: (V1) to the 13 month follow-up visit
Population: Intention to treat (ITT) sample. Multiple imputation with 8 datasets imputed via Markov Chain Monte Carlo sampling was used to handle missing data.
Measure: Mean (Standard Error); unit: weighted increment units/13 months
Groups:
- Placebo: Participants received a placebo dental coating containing no chlorhexidine diacetate (CHX).
- Active: Participants received a dental coating containing chlorhexidine diacetate (CHX) 10% weight per volume.
Arm/Group | Placebo | Active
Number analyzed (Participants) | 493 | 490
weighted increment units/13 months | 2.43 (0.32) | 2.68 (0.32)
Statistical Analysis 1: Comparison: Placebo vs Active; We hypothesized a lower increment score for the active treatment group but carried out two-tailed hypothesis testing. Sample size was estimated with simulated data with rank normalized scores. We calculated that 832 participants would yield a power of 90% to detect a 20% reduction in caries incidence (from a hypothesized mean increment of 1.5), and adopted a target of 1000 randomized participants to allow for attrition; Test type: Superiority or Other; p = 0.56, Regression, Linear — No interim analyses were done and no adjustment made for multiple comparisons. Identical analyses were run on each imputed dataset, with results combined with SAS® PROC MIANALZE to obtain final p-values; The primary outcome analysis included treatment and site as class variables and age and age-squared as continuous covariates; Mean Difference (Net) = 0.25, 95% CI 2-sided [-0.60 to 1.11], Standard Error of Mean 0.44

2. Secondary Outcome: Cumulative Net D12FS Caries Increment
Description: This measure was computed similar to the total net D12FS increment, but separately scored and combined transitions from the baseline to 7-month visits and from the 7- to 13-month visits, rather than simply looking at the baseline to 13-month visits.
Time Frame: Visit 1, 7-month follow-up, 13-month follow-up
Population: Intention-to-Treat sample
Measure: Mean (Standard Error); unit: caries increment units/13 months
Arm/Group | Placebo Dental Coating | Active Dental Coating (CHX)
Number analyzed (Participants) | 493 | 490
caries increment units/13 months | 5.53 (0.42) | 5.88 (0.43)
Statistical Analysis 1: Comparison: Placebo Dental Coating vs Active Dental Coating (CHX); hypothesized a reduced caries increment in active arm, though conducted two-tailed hypothesis test; Test type: Superiority or Other; p = 0.54, Regression, Linear — No adjustment for multiple comparisons. Identical analyses were run on each imputed dataset, with results combined with SAS® PROC MIANALYZE to obtain final p-values; Model included treatment and site as class variables and age and age-squared as continuous covariates; Mean Difference (Net) = 0.35, 95% CI 2-sided [-0.77 to 1.46], Standard Error of Mean 0.57

3. Secondary Outcome: Total Crude D12FS Caries Increment
Description: Computed analogous to the total net D12FS caries increment, but ignoring reversals (essentially assigned them zero weight). Computed only using baseline to 13-month visit data.
Time Frame: V1-13-month follow-up
Population: Intention-to-Treat sample
Measure: Mean (Standard Error); unit: caries increment units/13 months
Arm/Group | Placebo Dental Coating | Active Dental Coating (CHX)
Number analyzed (Participants) | 493 | 490
caries increment units/13 months | 6.47 (0.27) | 5.96 (0.28)
Statistical Analysis 1: Comparison: Placebo Dental Coating vs Active Dental Coating (CHX); Hypothesized lower increment in active arm, though hypothesis testing was two-sided; Test type: Superiority or Other; p = 0.18, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; treatment and site included as class variables and age and age-squared as continuous covariates; Mean Difference (Net) = -0.51, 95% CI 2-sided [-1.25 to 0.23], Standard Error of Mean 0.38

4. Secondary Outcome: Cumulative Crude D12FS Caries Increment
Description: This is computed analogous to the cumulative net D12FS increment, but ignoring reversals by assigning them weights of zero.
Time Frame: Visit 1, 7-month follow-up, 13-month follow-up
Population: Intention-to-Treat sample
Measure: Mean (Standard Error); unit: caries increment units/13 months
Arm/Group | Placebo Dental Coating | Active Dental Coating (CHX)
Number analyzed (Participants) | 493 | 490
caries increment units/13 months | 11.39 (0.42) | 10.72 (0.43)
Statistical Analysis 1: Comparison: Placebo Dental Coating vs Active Dental Coating (CHX); Hypothesized a lower increment for active treatment arm, although hypothesis testing was two-sided; Test type: Superiority or Other; p = 0.24, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Model included treatment and site as class variables, and age and age-squared as continuous covariates; Mean Difference (Net) = -0.68, 95% CI 2-sided [-1.80 to 0.45], Standard Deviation 0.57

ADVERSE EVENTS:
Time Frame: Adverse events were reported at any time throughout the study and were systematically screened for at the 6-month and 1-year visit.
Description: Systematic assessment of adverse events evaluated during routine completion of standard questionnaire.
Arm/Group | Placebo | Active
Serious Adverse Events (participants affected / at risk) | 31/493 | 28/490
Other Adverse Events (participants affected / at risk) | 87/493 | 84/490
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=493) | Active (N=490)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis of male external genital organ (Infections and infestations) | 1 (1) | 0 (0)
Cerebral ventricle dilation (Nervous system disorders) | 1 (1) | 0 (0)
Cervical spine stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Exposure to communicable disease (Social circumstances) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastric bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 2 (2) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lung injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Rectal fistula repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary bladder excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=493) | Active (N=490)
Nasopharyngitis (Infections and infestations) | 43 (44) | 30 (31)
Pharmaceutical product complaint (Social circumstances) | 12 (12) | 28 (28)
Sensitivity of teeth (Gastrointestinal disorders) | 32 (36) | 26 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No